CLINICAL TRIAL: NCT01226004
Title: Multi-Institutional Registry for Prostate Cancer Radiosurgery. An IRB Approved Observational Trial
Brief Title: Multi-Institutional Registry for Prostate Cancer Radiosurgery
Acronym: RPCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RPCR, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: FRRA01
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer Early Risk Treated by Radiosurgery; Prostate Cancer Intermediate Risk Treated by Radiosurgery
Keywords: radiosurgery; prostate; cancer; early; intermediate; CyberKnife
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To address pertinent questions regarding the utilization of stereotactic Body Radiotherapy (SBRT) to treat prostate cancer. The Florida Robotic Radiosurgery Association (FRRA) launched the first registry for prostate cancer patients treated with SBRT. The registry is designed to track surrogate treatment endpoints including prostate specific antigen (PSA), international prostate symptom score (IPSS),sexual health in men (SHIM), and visual analogue scale (VAS) scores, in addition to physical and survival data. Utilizing an independent vendor (Advertek, Inc.) experienced with the design and implementation of similar electronic registries, FRRA developed a data collection tool that staff members with a basic medical background can use to register and upload pertinent patient data, requiring no more than 20 to 30 minutes per patient. Participating patients will be monitored in follow-up for three years, with analysis and publication of the results semi-annually.

DETAILED DESCRIPTION:
To address pertinent questions regarding the utilization of radiosurgery (SBRT) to treat prostate cancer. The Florida Robotic Radiosurgery Association (FRRA) launched the first registry for prostate cancer patients treated with SBRT.

The registry is designed to track surrogate treatment endpoints including PSA, IPSS, SHIM, QOL, Karnofsky Performance Status, VAS scores, urine and bowel health, in addition to physical and survival data. Utilizing an independent vendor (Advertek, Inc.) experienced with the design and implementation of similar electronic registries.

FRRA developed a data collection tool that staff members with a basic medical background can use to register and upload pertinent patient data requiring no more than 20 to 30 minutes per patient. Participating patients will be monitored in follow-up for three years, with analysis and publication of the results semi-annually.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosis of prostate cancer
* early or intermediate risk

Exclusion Criteria:

* high risk prostate cancer

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men over 18 who have early or intermediate risk prostate cancer and have chosen to undergo radiosurgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-07; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Treatment Outcomes | 5 years
  Measurement of surrogate outcomes including IPSS and SHIM scores
Treatment toxicity | 5 years
  urinary and rectal complications as well as sexual health
Assess biochemical disease free survival using PSA | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark L. Perman, MD, Principal Investigator — South Florida Radiation Oncology, LLC.
Locations (44):
- United States (44):
  - CyberKnife of Birmingham, Birmingham, Alabama
  - University of South Alabama-USA Mitchell Cancer Institute, Mobile, Alabama
  - Phoenix CyberKnife & Radiation Oncology Center, Phoenix, Arizona
  - California Cancer Care, Fresno, California
  - Newport Diagnostic Center, Newport Beach, California
  - Scripps Clinic Radiation Therapy Centers, San Diego, California
  - Skyline Radiation Oncology, Tustin, California
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Colorado CyberKnife, Lafayette, Colorado
  - Anova Cancer Care, Lone Tree, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - CyberKnife Center of Miami, Miami, Florida
  - Naples Radiation Oncology, Naples, Florida
  - Memorial Cancer Institute CyberKnife Center, Pembroke Pines, Florida
  - CyberKnife Center of South Florida in Stuart, Stuart, Florida
  - CyberKnife Centers of Tampa Bay, Tampa, Florida
  - WellStar Research Insititute, Marietta, Georgia
  - CyberKnife Center of Chicago, Elmhurst, Illinois
  - Illinois Cyberknife, Park Ridge, Illinois
  - Baptist Health, Lexington, Kentucky
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Montana Cancer Institute Foundation, Missoula, Montana
  - St. Elizabeth CyberKnife Center, Lincoln, Nebraska
  - Las Vegas CyberKnife, Henderson, Nevada
  - Reno CyberKnife, Reno, Nevada
  - Riverview Medical Center, Red Bank, New Jersey
  - United Health Services, Johnson City, New York
  - First Dayton Cancer Care, Kettering, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - Oklahoma CyberKnife, Tulsa, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Philadelphia CyberKnife, Havertown, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Austin CyberKnife, Austin, Texas
  - Premier Cancer Centers, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - St. Luke's Medical Center, Houston, Texas
  - The START Center for Cancer Care, San Antonio, Texas
  - Cyberknife of Texas at East Texas Medical Center, Tyler, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Spokane CyberKnife, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - St. Mary's Medical Center, Huntington, West Virginia